CLINICAL TRIAL: NCT06205498
Title: Acalabrutinib Real World Italian obSErvational Secondary Data Collection Study of Acalabrutinib in the Treatment of Patients With Chronic Lymphocytic Leukemia.
Brief Title: Acalabrutinib Real World Italian obSErvational Study -ARISE
Acronym: ARISE
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Yghea (Unknown)
Responsible Party: Sponsor
Other Study IDs: D8221R00002
Record Dates: First submitted 2023-07-06; First posted 2024-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; acalabrutinib; CLL; Observational
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Drug: acalabrutinib — patients with CLL who initiated treatment with acalabrutinib over the period between 1st May 2021 and 30th April 2022, according to Italian legislation dlg 219/2006 art.125
  Other Names: Calquence

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common form of leukemia in the adults in the Western world, with an annual incidence of approximately 5 cases per 100,000 inhabitants in Italy.

Acalabrutinib (CalquenceTM), a selective second-generation Bruton Tyrosine Kinase (BTK) inhibitor developed by AstraZeneca, has been assessed for the treatment of CLL in three phase III clinical trials, ELEVATE-TN (treatment-naïve CLL), ASCEND and ELEVATE R/R (relapsed and refractory CLL). These pivotal randomized clinical trials established the efficacy and safety of acalabrutinib in patients with CLL and based on these data CalquenceTM received EMA approval in November 2020 for the treatment of CLL in adult patients and received AIFA (Agenzia Italiana del Farmaco) reimbursement as monotherapy in December 2021. However, further data are still required to evaluate the use of acalabrutinib in the real-life conditions of post-marketing authorization.

The primary aim of ARISE study is to evaluate the time to treatment discontinuation and reasons for discontinuation for acalabrutinib in a real world setting of patients with CLL. This study will provide the first real-world data on the use of acalabrutinib in the treatment of CLL in Italy.

DETAILED DESCRIPTION:
Study design:

This is an Italian non-interventional / observational, multicenter, longitudinal secondary data usage study based on a retrospective cohort of patients with CLL, who initiated treatment with acalabrutinib between 1st May 2021 and 30th April 2022 (index date), regardless of the treatment status at the time of inclusion. Each patient will be followed-up up to 5 years since the last enrolled patient index date (therefore for a maximum of 72 months). Five data extraction timepoints are planned for the investigators to proceed with secondary data extraction from patients' medical records and data entry into the electronic case report form (eCRFs).

Data Source(s):

Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time as part of patients' path of care (e.g., patient's hospital records, pharmacy dispensing records).

A standardized, validated eCRF will be developed to capture data extracted from source documents at each participating site.

Study Population:

All consecutive adult patients with CLL who initiated treatment with acalabrutinib over the period between 1st May 2021 and 30th April 2022, according to Italian legislation dlg 219/2006 art.125.

Outcome(s):

The primary outcome is the time to acalabrutinib discontinuation (defined as time in days from start date of acalabrutinib treatment to end date of acalabrutinib treatment).

Secondary outcomes include: Time from diagnosis to start of acalabrutinib, immunophenotype, CLL clinical stage (Binet), FISH profile, mutations, karyotype, CLL treatments before acalabrutinib, socio-demographic characteristics at baseline, medical history, concomitant treatments, COVID-19 prophylaxis and treatments, constitutional symptoms, patient clinical status, ECG/TTE, complete blood count with differential, serum chemistry, HIV and Hepatitis serology, active haemolysis, time to acalabrutinib discontinuation, acalabrutinib treatment (dosage, relative changes, temporary interruption/permanent discontinuation).

Exploratory outcomes include: Time to progression, Time to death, CLL status (according to iwCLL), Time to Next Treatment, Time to progression on next line treatment, reasons for ending of CLL treatments following acalabrutinib discontinuation, visits and hospitalizations due to CLL or suspected ADR during acalabrutinib treatment.

ELIGIBILITY:
Inclusion Criteria All consecutive patients with CLL who received acalabrutinib according to Italian legislation dlg 219/2006 art.125 will be eligible for inclusion in the study, subject to site agreement and patient consent to participate.

Patients must meet the following criteria for study entry:

1. Age ≥ 18 years old at the date of consent subscription.
2. Diagnosis of CLL.
3. Treatment of CLL with acalabrutinib at physician's discretion initiated between 1st May 2021 and 30th April 2022.
4. Informed consent to participate in the study and privacy form signed by the patient (or their legal representative).

Exclusion Criteria

Patients who meet any of the following criteria will be excluded:

1. Acalabrutinib treatment initiation before 1st May 2021 or after 30th April 2022.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators participating in this observational study should include all patients with CLL who initiated treatment with acalabrutinib over the period between May 1st, 2021 and April 30th, 2022, regardless of the treatment status at the time of inclusion. Thus, at the time of enrolment and retrospective data collection, patients may still be on treatment or have stopped treatment for any reason.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
time to acalabrutinib discontinuation | through study completion, an average of 5 years
  The primary outcome is the time to acalabrutinib discontinuation (defined as time in days from start date of acalabrutinib treatment to end date of acalabrutinib treatment) Kaplan-Meier median time to acalabrutinib discontinuation (defined as time in days from start date of acalabrutinib treatment to end date of acalabrutinib treatment).
  (Note: Any acalabrutinib treatment suspension >28 days is defined as discontinuation.
  Any acalabrutinib treatment suspension ≤ 28 days is defined as interruption and should not be considered for the analysis of the primary objective.

SECONDARY OUTCOMES:
demographic and clinical characteristics of CLL patients treated with acalabrutinib | baseline
  To describe demographic and clinical characteristics of CLL patients treated with acalabrutinib, by treatment line and potential associations with acalabrutinib permanent discontinuation.
describe acalabrutinib treatment patterns | through study completion, an average of 5 years
  Duration of acalabrutinib suspension= time from the date of last dose before suspension to the date of acalabrutinib restart.
  Frequency of acalabrutinib interruptions Time to interruption= time from the first dose of acalabrutinib to the date of last dose before interruption Proportion of each reason for treatment ending (adverse events, disease progression, compliance issues, patient's decision, physician's choice, death, other) In case of discontinuation for adverse event: proportion of each type of adverse event.
  Frequency of acalabrutinib dose changes Proportion of each reason for dose change Time to dose change= time from the first dose of acalabrutinib to the first dose administered at the new dosage Mean dose at last acalabrutinib use Relative dose intensity= received dose/prescribed dose (where received dose is the total dose actually received by patient during the whole observation period; prescribed dose is the dose at the acalabrutinib )initiation
CLL clinical stage | baseline
  according to Binet staging system (stage A, B, C) according to Eichhorst et al., 2020.
FISH profile | baseline
  del(11q) del(17p); trisomy 12; del(13q); normal
Date of birth | baseline
  month/year
gender | baseline
  male or famale
Height | baseline
  cm
Weight | throught study completion, an average of 5 years
  Kg
Body Mass Index | Through study completion, an average of 5 years
  kg/m2
Medical illness burden | Through study completion, an average of 5 years
  CIRS-G scale
Red blood cell count | Through study completion, an average of 5 years
  x10^12/L
White blood cell count | Through study completion, an average of 5 years
  x10^9/L
platelets count | Through study completion, an average of 5 years
  x10^9/L
hemoglobin | Through study completion, an average of 5 years
  gr/dL
differential count of lymphocytes and neutrophils | Through study completion, an average of 5 years
creatinine clearance (mL/min), aspartate transaminase (AST; U/L), alanine transaminase (ALT; U/L), gamma-glutamyl transferase (GGT; U/L), bilirubin (mg/dL), LDH (U/L), β2-microglobulin (mg/dL), IgG, IgA, IgM levels (mg/dL) | baseline
Anti-HIV antibodies test and Hepatitis serology tests including hepatitis B surface antigen (HbsAg), hepatitis B surface antibody (HbsAb), hepatitis B core antibody (anti-HBc), and hepatitis C (HCV) antibody | baseline

OTHER OUTCOMES:
measure effectiveness of acalabrutinib | through study completion, an average of 5 years
  To measure effectiveness of acalabrutinib treatment in patients with CLL in terms of:
  Progression Free Survival (PFS), Overall Survival (OS), Overall Response Rate (ORR - categorization according to iwCLL), Time To Next Treatment (TTNT) Kaplan-Meier median time to progression (defined as time from start date of acalabrutinib treatment to the first assessment of disease progression) Kaplan-Meier median time to Death (defined as time from start date of acalabrutinib treatment to death) Proportion of patients with Complete Response, Partial response, Partial Response with lymphocytosis or Stable Disease Kaplan-Meier median time to next treatment (defined as time from start date of acalabrutinib treatment to the first consecutive treatment)
evaluate effectiveness of CLL treatments following acalabrutinib discontinuation | through study completion, an average of 5 years
  To evaluate effectiveness of CLL treatments following acalabrutinib discontinuation in terms of PFS2, OS and ORR by treatment and relative causes of discontinuation.
  Kaplan-Meier median time to progression (defined as time from start date of acalabrutinib treatment to progression) on next-line treatment The time to death and the overall response are computed as described for the exploratory objective n.1 Proportion of each reason for discontinuation of CLL treatments following acalabrutinib (patient's decision, physician's choice, adverse events, death, other, unknown)
estimate Healthcare Resources Utilization | through study completion, an average of 5 years
  To estimate Healthcare Resources Utilization by patients with CLL, in terms of hospitalizations and visits (routine follow-up, outpatient visits and emergency visits) Total visits= number of all visits performed during the observation period Total hospitalizations= number of all hospitalizations performed during the observation period Mean, minimum and maximum total visits Mean, minimum and maximum total hospitalizations Mean, minimum and maximum hospitalizations duration In case of visits and hospitalization due to AE suspected of relationship with acalabrutinib (ADR): proportion of each type of adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Carola Boccomini, Principal Investigator — AOU Città della Salute e della Scienza di Torino - Presidio Molinette; Chiara Borrella, Principal Investigator — IRCCS San Gerardo Monza; Catello Califano, Principal Investigator — PO A. TORTORA; Daniele Caracciolo, Principal Investigator — AOU Mater Domini / Università Magna Grecia; Gioacchino Catania, Principal Investigator — AO SS Antonio e Biagio e Cesare Arrigo; Marta Coscia, Principal Investigator — AOU Città della Salute e della Scienza; Luigi Curreli, Principal Investigator — PO San Martino; Giovanni D'Arena, Principal Investigator — PO S.Luca - DEA I livello; Federica De Marco, Principal Investigator — Ospedale San Giovanni Bosco, ASL Città di Torino; Gaetano De Santis, Principal Investigator — Ospedale "Mon. Dimiccoli" Barletta; Nicola Di Renzo, Principal Investigator — PO Vito Fazzi ASL di Lecce; Ambra Di Veroli, Principal Investigator — ASL Viterbo; Amalia Stefania Figuera, Principal Investigator — AOU Policlinico G.Rodolico - San Marco; Myriam Foglietta, Principal Investigator — AO S. Croce e Carle; Vincenzo Fraticelli, Principal Investigator — Responsible Research Hospital; Susanna Gallo, Principal Investigator — ASLTO4 Sedi di Ciriè - Chivasso ed Ivrea; Massimo Gentile, Principal Investigator — AO Cosenza; Giulio Giordano, Principal Investigator — Ospedale di riferimento regionale "A. Cardarelli" - Campobasso; Adalberto Ibatici, Principal Investigator — Ospedale Policlinico San Martino; Luca Laurenti, Principal Investigator — Policlinico Universitario Gemelli IRCCS; Massimo Magagnoli, Principal Investigator — Istituto Clinico Humanitas; Luigi Malandruccolo, Principal Investigator — Ospedale Spaziani - ASL Frosinone; Alessandro Noto, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Francesca Romana Mauro, Principal Investigator — Università Sapienza di Roma; Carla Minoia, Principal Investigator — IRCCS Giovanni Paolo II; Roberta Murru, Principal Investigator — Ospedale Oncologico" A. Businco" - ARNAS "G. Brotzu"; Marina Motta, Principal Investigator — Asst Degli Spedali Civili Di Brescia; Pellegrino Musto, Principal Investigator — AOU Policlinico Consorziale di Bari; Marco De Gobbi, Principal Investigator — AOU San Luigi Gonzaga; Getano Palumbo, Principal Investigator — Ospedali Riuniti di Foggia; Fabrizio Pane, Principal Investigator — Federico II University; Maria Cristina Pasquini, Principal Investigator — Ospedale Maggiore Crema; Domenico Pastore, Principal Investigator — PO "A.Perrino" di Brindisi; Elsa Pennese, Principal Investigator — ASL Pescara; Rosario Potito Scalzulli, Principal Investigator — IRCCS Casa Sollievo della Sofferenza; Lydia Scarfò, Principal Investigator — IRCCS Ospedale San Raffaele; Ilaria Scortechini, Principal Investigator — AOU delle Marche; Paolo Sportoletti, Principal Investigator — Università degli Studi di Perugia - Azienda Ospedaliera S.M. Perugia; Caterina Cecilia Stelitano, Principal Investigator — Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli; Agostino Tafuri, Principal Investigator — AOU Sant'Andrea; Anna Tamburini, Principal Investigator — Azienda Ospedaliera S. Giovanni Addolorata; Monica Tani, Principal Investigator — Ospedale Santa Maria delle Croci - Ravenna; Vincenzo Pavone, Principal Investigator — Azienda Ospedaliera Cardinale G. Panico; Andrea Visentin, Principal Investigator — Azienda Ospedale Università Padova; Massimiliano Postorino, Principal Investigator — Ospedale Policlinico Tor Vergata; Laura Nocilli, Principal Investigator — Ospedale Papardo
Locations (33):
- Italy (33):
  - Research Site, Alessandria
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Barletta
  - Research Site, Brindisi
  - Research Site, Campobasso
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Cosenza
  - Research Site, Crema
  - Research Site, Cuneo
  - Research Site, Foggia
  - Research Site, Frosinone
  - Research Site, Genova
  - Research Site, Lecce
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pagani
  - Research Site, Perugia
  - Research Site, Pescara
  - Research Site, Ravenna
  - Research Site, Reggio Calabria
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Salerno
  - Research Site, San Giovanni Rotondo
  - Research Site, Torino
  - Research Site, Tricase
  - Research Site, Varese
  - Research Site, Viterbo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/